CLINICAL TRIAL: NCT06943963
Title: The Effect of Self Stigma Tailored Cognitive Behavioral Therapy on Gambling Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ayça Çınaroğlu Asar, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-3.1/60
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Results first posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Gambling Addiction; Gambling Disorder; Gambling Disorder Treatment; Stigma; Stigma of Mental Illness; Self Stigma; CBT; Cognitive Behavioral Therapy
Keywords: self stigma; CBT; gambling disorder; gambling addiction; controlled trial; therapy
MeSH Terms: conditions — Gambling; Social Stigma

STUDY DESIGN:
Intervention Model Description: This study uses a randomized controlled trial design with an intervention and control group. Participants diagnosed with Gambling Disorder and followed at the Ege University Institute of Substance Addiction, Toxicology and Pharmaceutical Sciences were randomly assigned to the intervention or control group.The intervention group underwent a four-session structured cognitive behavioral therapy (CBT) program specifically designed to address self-stigma, while the control group received treatment as usual.Pre- and post-test assessments were conducted using the Self-Stigma Scale (SSS) and the South Oaks Gambling Screen (SOGS) to assess changes in self-stigma perception and gambling severity. Additionally, a follow-up assessment was conducted one month after post-testing to measure sustainability of improvements over time. A power analysis determined that 26 participants (13 per group) were required for a power of 0.80. To account for potential dropouts, the sample size was increased by 20%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Intervention) Group (Experimental): Participants in the research arm received "Self Stigma Tailored Cognitive Behavioral Therapy on Gambling Disorder" addition to the standard treatment for Gambling Disorder (GD) provided at the Addiction Clinic.
  The standard treatment includes the medical treatment for GD and motivational interviews administered by a psychiatrist at the Addiction Clinic where the research is conducted.
  Interventions: Behavioral: Self Stigma Tailored Cognitive Behavioral Therapy on Gambling Disorder; Drug: standart pharmacotherapy; Behavioral: motivational intervention
- Control Group (Active Comparator): Participants in the control group received the standard treatment for Gambling Disorder (GD), as described in the previous paragraph, at the Institute's Addiction Clinic. The duration and type of treatment were tailored to the individual patient by the psychiatrist. During the period when the experimental group received the Self Stigma Tailored Cognitive Behavioral Therapy for Gambling Disorder, the control group participants were placed on the waiting list and did not receive any specific intervention for self-stigma perception.
  Interventions: Drug: standart pharmacotherapy; Behavioral: motivational intervention

INTERVENTIONS:
Behavioral: Self Stigma Tailored Cognitive Behavioral Therapy on Gambling Disorder — The Self Stigma Tailored Cognitive Behavioral Therapy for Gambling Disorder (SSCBT) is a novel intervention designed specifically for this study and has not been previously used or named in existing literature. This 4-session protocol can be integrated into any part of GD treatment. Each session was accompanied by materials specifically designed for that session's content, and assignments related to the session's topics were given at the end of each session.
  Session 1: Gambling Disorder from a bio-psycho-social perspective, stigma and self-stigma, CBT introduction, cognitive-behavioral model of self-stigmatization, impact of emotions and cognitive distortions.
  S. 2: Self-stigmatizing thoughts and behaviors, identifying automatic thoughts with cognitive techniques, cognitive awareness, and restructuring with evidence examination.
  S. 3: Aligning behaviors with values, cognitive restructuring, behavior change, and self-awareness.
  S. 4: Prevention strategies, relapse prevention planning.
  Other Names: SSCBT
  Arms: Experimental (Intervention) Group
Drug: standart pharmacotherapy — All participants continued to receive standard pharmacotherapy from their respective psychiatrists.
Behavioral: motivational intervention — All participants continued to receive the standard motivational interviewing intervention for addiction from their psychiatrist.

SUMMARY:
The goal of this clinical trial was to evaluate whether a cognitive behavioral therapy (CBT) program focused on self-stigma could help reduce both self-stigma and gambling disorder severity in adults diagnosed with gambling disorder.

The main questions it aimed to answer were:

Did self-stigma-focused CBT lower self-stigmatizing thoughts in individuals with gambling disorder? Did the severity of gambling disorder symptoms decrease after the intervention? Did these changes remain stable after the treatment ended? Did self-stigma play a role in how the treatment worked? Participants were assigned to either an intervention group or a control group. Completed assessments before the treatment, after the treatment, and during the 1 month follow-up period.

Participants in the intervention group:

Received four sessions of cognitive behavioral therapy (face-to-face or online) targeting self-stigmatizing thoughts related to gambling Researchers compared the intervention and control groups to observe whether self-stigmatization affected treatment outcomes. Surveys used in this study included a self-stigma scale and the South Oaks Gambling Screen (SOGS).

A total of 26 participants (13 in each group) were enrolled in the study; in addition, 3 extra participants per group were included to account for possible dropouts.

The results were analyzed using statistical methods.

DETAILED DESCRIPTION:
The total duration of the study is 13 months, from March 2024 to April 2025. The stages of the study were planned according to weeks (W). The timeline and phases of the study are as follows:

1. Sample screening - March 2024, W1-W4
2. Assessment session and pre-test measurements (March 2024, W2-W4)
3. Randomization and assignment of research groups (April 2024, W5-W6)
4. Informing the participants (April 2024, W5-W6)
5. Intervention (psychotherapy sessions) (April 2024 - September 2024, W7-W20)
6. Post-test measurements (September 2024 - October 2024, W21-W23)
7. Follow-up measurements (December 2024 - January 2025, W27-W29)
8. Data analysis (January 2025, W30-W32)
9. Reporting (February 2025 - April 2025, W33-W39)

<!-- -->

1. Sample Screening Face-to-face or telephone interviews were conducted with patients who applied to the Addiction Unit of the Institute on Drug Abuse, Toxicology and Pharmaceutical Sciences at Ege University. For patients diagnosed with Gambling Disorder at the outpatient clinic, appointments were scheduled for face-to-face assessments. Preliminary interviews and appointment scheduling continued until a sufficient number of participants were reached.
2. Assessment Session and Pre-Test Measurements

   The steps of the assessment session (clinical evaluation) are as follows:

   • Providing detailed information about the study to patients who participated in the assessment session.
   * Informing the participants that they would be randomly assigned to one of two groups through a randomization program by a researcher other than the primary investigator.
   * Obtaining signed informed consent forms from patients who voluntarily agreed to participate in the study, and providing them with a copy.
   * Taking the anamnesis of patients who agreed to participate voluntarily. Anamnesis information was recorded in the Case Report Form developed by the principal investigator.
   * Administering all scales (Self-Stigma Scale and South Oaks Gambling Screen) to participants with the guidance of the principal investigator. These measurements constitute the baseline (t0) assessments of the study.
   * Informing the participants that they would be contacted again to be informed about their group assignment before the session ends.
3. Randomization and Research Groups Participants were stratified based on their Self-Stigma Scale scores using the SPSS program, and then randomly assigned to the intervention and control groups within each stratum. To prevent selection bias, the random assignment of participants to groups was performed by a different researcher.
4. Informing the Participants After group assignment, participants in the intervention group were contacted to schedule their first psychotherapy session. Participants in the control group were informed that they had been placed on a waitlist. Patients who were found to be ineligible for participation based on exclusion criteria were also contacted and informed that they would not be included in the study.
5. Intervention (Psychotherapy Sessions): Self-Stigma Tailored Cognitive Behavioral Therapy on Gambling Disorder (SSCBT-GD) The SSCBT-GD intervention will be conducted with participants in the intervention group according to a structured protocol, scheduled at mutually agreed dates and times. Each psychotherapy session will be conducted approximately one week apart. The duration of each session is 60 minutes. The intervention consists of a total of four sessions, unless otherwise interrupted (e.g., participant rescheduling a session).

   Intervention Plan:

   Session 1: Psychoeducation I • Addressing Gambling Disorder from a bio-psycho-social perspective.
   * Explaining the concepts of social stigma and self-stigma.
   * Providing information on Cognitive Behavioral Therapy (CBT).
   * Presenting the cognitive-behavioral model related to self-stigmatization in individuals with Gambling Disorder.
   * Exploring the impact of emotions and cognitive distortions.

   Materials:

   Operant learning model of Gambling Disorder, progressive model of stigma, progressive model of self-stigma, bio-psycho-social CBT model.

   Session 2: Psychoeducation II

   • Examining self-stigmatizing thoughts and their impact on behavior.

   • Identifying automatic thoughts relevant to the individual's symptoms using cognitive techniques.

   • Introducing cognitive awareness and the foundations of cognitive restructuring through evidence-based examination techniques.

   Materials:

   Emotion-thought-behavior connection, thought and emotion analysis, evidence vs. counter-evidence examples and practice, thought-emotion reevaluation.

   Session 3: Psychoeducation III • Aligning behaviors with personal values.

   • Addressing goals for cognitive restructuring and behavioral change.

   • Enhancing self-awareness.

   Materials:

   Values model, summary reminder, vicious cycle diagram.

   Session 4: Psychoeducation IV • Exploring the interaction between emotions, thoughts, and behaviors. • Increasing awareness of personal life patterns and experiences. • Discussing foresight and preventative strategies.

   • Relapse prevention strategies and termination process.

   Materials:

   Integrated summary of addiction and self-stigma, example triggering thoughts, relapse prevention form.

   Homework Assignments Homework is a technique commonly used in CBT interventions to reinforce therapeutic gains. Its goal is to support participants in internalizing the intervention content by engaging with the material between sessions. These assignments remain with the participant and serve as a summary of their therapeutic journey.

   • Homework 1: Problem List - Aims to assess the participant's current awareness of the problem.

   • Homework 2: A-B-C (Illustrated) - Helps recognize and label thoughts and emotions in specific situations.

   • Homework 3: New Book, Old Book - Encourages the participant to explore emotions, thoughts, and alternative perspectives.
   * Homework 4: Behavioral Experiment Form - Offers an opportunity to challenge and restructure personal cognitions through practical exercises.
   * Homework 5: Relapse Prevention Form - Assists in documenting new experiences and serves as a reminder of session content during the cognitive restructuring phase.

   Participants who attended only one, two, or three psychotherapy sessions were not considered to have completed the intervention. Only those who participated in all four sessions were deemed to have completed it.

   Treatment as Usual (TAU):

   Throughout the SSCBT-GD intervention, all participants in both the experimental and control groups continued to receive TAU from the addiction outpatient clinic. The content and duration of TAU were determined individually by the clinic psychiatrist. TAU primarily consisted of medical treatment and motivational interviewing when necessary.
6. Post-Intervention and Follow-Up Assessments The Self-Stigma Scale and South Oaks Gambling Screen were used as measurement tools for both post-intervention and follow-up assessments. These assessments were conducted simultaneously for participants in both the experimental and control groups.

   Post-intervention assessments (t1) were conducted four weeks after the start of the intervention (the date of the first psychotherapy session was considered the start date).

   Follow-up assessments (t2) were conducted four weeks after the post-intervention assessments.
7. Data Analysis After the follow-up assessments were completed, the data collected through the measurement tools were analyzed. The experimental and control groups were compared in terms of the study's dependent variables.
8. Intervention for the Control Group If the analysis revealed that participants in the experimental group benefited from the SSCBT-GD intervention, the same intervention was offered to the control group for ethical reasons
9. Reporting The research process and findings were documented and presented in tabular format. The reporting phase constituted the final stage of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the diagnostic criteria for Gambling Disorder (GD) according to the DSM-5:
2. Currently receiving or having completed the standard treatment provided at the outpatient clinic.
3. Scoring 72 or above on the Self Stigma Scale.
4. Being between 18 and 65 years old.

Exclusion Criteria:

1. "Intellectual Disability" classified under neurodevelopmental disorders.
2. "Communication Disorders" resulting from neurodevelopmental disorders or another medical condition.
3. Based on clinical interviews and DSM-5 diagnostic criteria:
4. "Bipolar and Related Disorders" with psychotic features.
5. "Depressive Disorders" with psychotic features.
6. "Dissociative Disorders" such as depersonalization, derealization, or identity disruption.
7. Any disorder classified under "Schizophrenia Spectrum and Other Psychotic Disorders," including schizophrenia, schizotypal personality disorder, and schizoaffective disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Umut Kırlı, Assoc. Prof., Study Director — Ege University, Addiction Clinic within the Institute of Addiction, Toxicology, and Pharmaceutical Sciences.; Ayça Çınaroğlu Asar, B.A., Principal Investigator
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
As the study has not yet been published, the plan to share individual participant data (IPD) is to be determined after the publication of the results.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: "Participants were recruited from the Addiction Unit of the Institute on Drug Abuse, Toxicology and Pharmaceutical Sciences at Ege University between March 2024 and April 2025. Recruitment involved face-to-face and telephone screening of patients diagnosed with Gambling Disorder during routine outpatient admissions. Screening continued until the required sample size was reached.
Pre-assignment Details: Records of 66 patients were screened. Eleven did not meet criteria. Of the remaining 55, two lived outside the city, 13 could not be reached, and five declined. Thirty-five attended baseline assessment; nine were excluded due to low Self-Stigma scores. In total, 26 eligible participants were enrolled and randomized.
Period: Overall Study
Arm/Group | Experimental (Intervention) Group | Control Group
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analyses included only participants who met the predefined eligibility criteria for the study: having a current diagnosis of Gambling Disorder and scoring 72 or above on the Self-Stigma Scale at baseline (T0). Participants who did not meet these criteria or had incomplete baseline assessments were excluded from the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental (Intervention) Group | Control Group | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] — Age (years) was recorded for each participant using the case report form at baseline. Each participant reported their own age at the time of enrollment.
  years | 36.5 (9.77) | 30 (4.8) | 33.25 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex was recorded for each participant using the case report form at baseline.
  Participants
    Female | 0 | 2 | 2
    Male | 13 | 11 | 24
Self-Stigma Scale [Mean (Standard Deviation); unit: self stigma scale score] — Self-stigmatization related to gambling disorder, assessed using the Self-Stigma Scale (SSS), a self-report questionnaire consisting of 36 items (in Turkish version) rated on a Likert-type scale. Total scores range from 36 to 144, with higher scores indicating greater levels of internalized stigma. Baseline assessment was conducted prior to the intervention. Participants scoring above 72 were included in the study.
  self stigma scale score | 118.15 (13) | 113.31 (13) | 115.73 (13)
South Oaks Gambling Screen [Mean (Standard Deviation); unit: South Oaks Gamblin Screen Score] — Gambling severity, assessed using the South Oaks Gambling Screen (SOGS), a self-report screening instrument consisting of 19 items (Turkish version) designed to identify gambling-related problems. Total scores range from 0 to 19, with higher scores indicating greater severity of gambling problems. The scale was administered at baseline and repeated over time to assess changes in gambling severity across the study period. Baseline assessment was conducted prior to the intervention.
  South Oaks Gamblin Screen Score | 14.25 (2) | 10.85 (1.6) | 12.55 (1.83)
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Self-Stigmatization Score as Measured by the Self-Stigma Scale (SSS). Baseline (Week 0) to Post-treatment (Week 4) and Follow-up (Week 8)
Description: Self-stigma will be measured using the Self-Stigma Scale (SSS). Scores range from 36 to 144, with 72 and higher scores indicating severe self-stigmatization. Changes from baseline (Week0) to post-treatment (Week 4) and follow-up (Week 8) will be analyzed.
Time Frame: post-treatment (Week 4) and follow-up (Week 8)
Measure: Mean (Standard Deviation); unit: Self Stigma Scale Scores
Arm/Group | Experimental (Intervention) Group | Control Group
Number analyzed (Participants) | 13 | 13
Self Stigma Scale Scores
  post intervention (t1) | 82.77 (24.43) | 110.3 (17)
  follow up (t2) | 80.38 (21.25) | 105.92 (18.78)
Statistical Analysis 1: Comparison: Experimental (Intervention) Group vs Control Group; A mixed-design ANOVA was used to compare repeated measurements of the dependent variables across groups. To examine changes in the dependent variables over time between groups, the interaction between the independent variable and time (group × time) was analyzed; Test type: Other — Repeated measures/Mixed-Design ANOVA; p < 0.05, ANOVA; Mean Difference (Net) = 0.002; F value (from ANOVA): 6.30

2. Primary Outcome: Change in Gambling Severity Score as Measured by the South Oaks Gambling Screen (SOGS). Baseline (Week 0) to Post-treatment (Week 4) and Follow-up (Week 8)
Description: Gambling severity will be assessed using the South Oaks Gambling Screen (SOGS). Scores range from 0 to 19, with higher scores indicating greater gambling-related problems. Changes from baseline to post-treatment and follow-up will be analyzed.
Time Frame: post-treatment (Week 4) and follow-up (Week 8)
Measure: Mean (Standard Deviation); unit: South Oaks Gambling Screen Scores
Arm/Group | Experimental (Intervention) Group | Control Group
Number analyzed (Participants) | 13 | 13
South Oaks Gambling Screen Scores
  post intervention (t1) | 3.77 (1.96) | 7.38 (4.19)
  follow up (t2) | 4.46 (2.87) | 5.31 (2.62)
Statistical Analysis 1: Comparison: Experimental (Intervention) Group vs Control Group; Test type: Other — Repeated Measures/ Mixed Design ANOVA; p < 0.05, ANOVA; Mean Difference (Net) = 0.0001; F value (from ANOVA): 10.75

3. Post Hoc Outcome: Mediation Analyze
Description: Mediation analysis was conducted to examine whether [Self Stigma score change, M] mediates the effect of [being intervention group or control group, X] on [south oaks gambling screen score change, Y]. Change scores from baseline (week 0) to post-intervention (week 4) (t1 - t0) were used in the analysis. Used Process Macro Model 4.
Time Frame: Outcome measures at post-intervention (after the fourth session, week 4; T1) were compared to baseline scores (prior to intervention; T0) by calculating change scores as T1 minus T0.
Measure: Number (95% Confidence Interval); unit: beta coefficient -Scores Changes (t1-t0)
Groups:
- All Participants: mediation analysis was conducted with all participants to examine whether change in Self-Stigma (Mediator, M) mediates the effect of intervention group (X) on change in gambling severity (Y). Change scores from baseline to post-intervention (t1 - t0) were used.
  X = group (experiment vs control) M = Self-Stigma score means changes Y = SOGS score means changes
Arm/Group | All Participants
Number analyzed (Participants) | 26
beta coefficient -Scores Changes (t1-t0)
  Direct Effect X= group type (intervention or control) to Y= SOGS scores changes | -2.11 [-5.17 to 0.94]
  X= group type (intervention or control) to M= SSS score changes | -32.38 [-45.93 to -18.83]
  M= SSS score changes to Y= SOGS scores changes | 0.14 [0.08 to 0.21]

ADVERSE EVENTS:
Time Frame: from baseline measures until end of follow up, up to 8 weeks
Description: Adverse events were monitored informally through participant self-report and therapist observation during the intervention period. No serious adverse events were anticipated or observed in this behavioral intervention study.
Arm/Group | Experimental (Intervention) Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
The groups were not fully balanced in baseline gambling severity, which may influence interpretation of the results. The study was not placebo-controlled or blinded, which could affect participant responses. Additionally, the one-month follow-up limits conclusions about the long-term effects of the intervention.Since SSCBT is a newly developed intervention model, further studies with larger and more diverse samples are needed to strengthen the evidence base.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-12-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT06943963/Prot_SAP_ICF_001.pdf